CLINICAL TRIAL: NCT04983433
Title: Increasing Amyloidosis Awareness and Diagnosis Through Programmatic Imaging, Blood/Urine Testing and Pathology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Principal Investigator, Dr Phillip Scheinberg, Head of Hematology, Beneficência Portuguesa de São Paulo
Other Study IDs: Amyloidosis
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-07

CONDITIONS: Amyloidosis
Keywords: Amyloid cardiomyopathy
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To set up a Brazilian strategy for early diagnosis of cardiac amyloidosis using new modality of echocardiography, the 3D echocardiography, and the level of myocardial deformity by measuring the Strain Longitudinal through the technology Speckle Tracking.

DETAILED DESCRIPTION:
Transthyretin cardiac amyloidosis (ATTR-CA) is an infiltrative cardiomyopathy caused by extracellular deposition of insoluble transthyretin amyloid fibrils in the myocardium. Unstable changes in the wild type and variant (familial) stimulate misfold aggregation and ultimately form amyloid fibrils and deposit in various tissues including the heart. Generally, cardiac amyloidosis is a cause of heart failure with preserved ejection fraction. The heart involvement with amyloidosis may represent part of a systemic disease with multiorgan involvement as is seen with light chain amyloidosis (AL). A distinct form of cardiac amyloidosis is the deposition of misfold transthyretin that results from aggregation of the native protein or from inherited mutations in the transthyreyin (TTR) gene, in particular in old patients and, with the increase of the aged population, the incidence of ATTR-CA is increasing although its real presence and correct diagnosis lacks standardized strategies, in particular due to diseases in the differential diagnosis with similar phenotypes. The Wild type ATTR-CA also known as senile systemic amyloidosis caused by age related misfolding of the TTR is the most frequent form of age-related cardiac amyloidosis. Hereditary ATTR-CA due to gene mutations can also lead to cardiac amyloidosis but in Brazil the most frequent mutation Val30Met usually has a clinical phenotype predominantly neurological contrary to the USA, where the mutation Val122Ile is more frequent with a cardiomyopathy phenotype. Lack of recognition of cardiac amyloidosis due to the presence of nonspecific symptoms and associated comorbidities commonly leads to delayed diagnosis and disease progression. Echocardiography is the first line technique for patients presenting with heart failure but there is still a gap on the clinical utility of the multiparametric parameters or their combination in patients where conventional echocardiogram raises the suspicion of cardiac amyloidosis. The study will be one of the first in its kind to prospectively delineate the presence of cardiac amyloidosis in a patient population where this hypothesis has not been properly evaluated.

Study Design:In this cohort study, patients undergoing evaluation for amyloidosis will be provided with diagnostic tools to confirm the diagnosis; in cases where verified, subtype methodologies for amyloidosis subtype characterization will be employed. If there is a suspicion of amyloidosis complementary imaging, etiologic evaluation with TTR sequencing, paraprotein evaluation (serum and urine serum protein electrophoresis and immunofixation, serum-free light), and pyrophosphate scintigraphy will be performed. If the origin of amyloid protein cannot be determined, further evaluation with biopsy of the amyloid deposition and mass spectrometry will be undertaken. Initially, fatpad biopsy and minor salivary glands will be performed. If unrevealing, the affected organ will be biopsied for amyloid tissue characterization.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with heart failure in the absence of hypertension
* heart failure with normal ejection fraction
* heart failure associated with aortic stenosis and atypical arrythmias, in which there is the suspicion of cardiaca amyloidosis

Exclusion Criteria:

* Individuals which do not consent to participate on the study or those that retired the consent during the study
* Individuals under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure in the aged population. Approximately 100 patients will be screened on the patient population described.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with diagnosis of ATTR cardiac amyloidosis after performing protocol exams (not necessarily all) - echocardiogram, cardiac magnetic resonance, scintigraphy, genetic test, blood and urine paraprotein test and biopsies. | After performing protocol exams, which will occur, for each patient, approximately, two months after entry in the study.
  Infiltrative cardiomyopathy caused by extracellular deposition of insoluble transthyretin amyloid fibrils in the myocardium.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Scheinberg, MD, Principal Investigator — Beneficência Portuguesa de São Paulo
Locations (1):
- Gisele Medeiros Bastos, São Paulo, São Paulo, Brazil